CLINICAL TRIAL: NCT00786331
Title: Randomized Phase II Study of Pemetrexed Versus Pemetrexed and Carboplatin as Second Line Chemotherapy in Advanced Non-small-cell Lung Cancer (NSCLC).
Brief Title: Pemetrexed +/- Carboplatin as Second Line Treatment in NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Responsible Party: Dr. Corrado Boni, GOIRC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOIRC 02/2006; EudraCT number 2006-004009-24
Record Dates: First submitted 2008-07-01; First posted 2008-11-06 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Advanced Non-Small Cell Lung Cancer
Keywords: second line treatment; pemetrexed; carboplatin
MeSH Terms: interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Monochemotherapy
  Interventions: Drug: Pemetrexed
- B (Experimental): Combination chemotherapy
  Interventions: Drug: Pemetrexed plus carboplatin

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed 500 mg/m2 i.v. over approximately 10 minutes on day 1 of a 21 days cycle
  Arms: A
Drug: Pemetrexed plus carboplatin — Pemetrexed 500 mg/m2 i.v. over approximately 10 minutes on day 1 and Carboplatin AUC 5 i.v. over approximately 30 minutes on day 1 (beginning approximately 30 minutes after the end of the pemetrexed infusion) of a 21 days cycle
  Arms: B

SUMMARY:
The aim of this study is to compare time to progression between the combination pemetrexed-carboplatin and pemetrexed alone in previously treated patients with locally advanced or metastatic NSCLC.

DETAILED DESCRIPTION:
In spite of the superiority of single agent over best supportive care in second-line NSCLC, the prognosis of these patients remains poor with a median survival of 6-7 months, justifying the evaluation of new regimens in this setting. An open question in the second-line treatment of NSCLC remains the possible superiority of combination chemotherapy over single agent, as it has been clearly demonstrated in first-line. Particularly, the addition of platinum to either docetaxel or pemetrexed should be further investigated especially in patients with prior response/stable disease to platinum-based first-line chemotherapy. Pemetrexed has shown anti-tumor activity in combination with other chemotherapy agents, including gemcitabine, vinorelbine, taxanes, cisplatin and carboplatin. In this multicenter, open label, randomized phase II trial, pemetrexed 500 mg/m2 and carboplatin AUC 5 will be administered on day 1 every 3 weeks until progression of disease or for a maximum of 4 courses in the experimental arm. The control arm will be pemetrexed as single agent at 500 mg/m2 on day 1 every 3 weeks until progression of disease or for a maximum of 4 courses.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* Histologically or cytologically confirmed non-small-cell lung cancer
* Unresectable stage IIIB, stage IV and unresectable local relapse or metastatic disease, with evidence of disease progression after first line chemotherapy which should have included a platinum agent.
* ECOG performance status lower than or equal to 2
* Adequate hematological, hepatic and renal functions
* Life expectancy greater than or equal to 12 weeks
* Prior treatment with only 1 chemotherapy regimen for the treatment of advanced disease which should have included a platinum agent
* At baseline, presence of at least one measurable target lesion as per RECIST criteria

Exclusion Criteria:

* Prior treatment with pemetrexed.
* Patients who are pregnant or lactating
* Patients with any underlying medical condition that might be aggravated by treatment or which cannot be controlled.
* Symptomatic brain metastases
* History of another malignancy within the past five years except basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Concomitant treatment with any other anticancer drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To compare time to progression between the combination pemetrexed-carboplatin and pemetrexed alone in previously treated patients with locally advanced or metastatic NSCLC | 36 months

SECONDARY OUTCOMES:
To assess differences in terms of response rate between the combination pemetrexed-carboplatin and pemetrexed alone. | 3 months
To assess differences in terms of duration of response between the combination pemetrexed-carboplatin and pemetrexed alone. | 36 months
To assess differences in terms of toxicity between the combination pemetrexed-carboplatin and pemetrexed alone. | 3 months
To assess differences in terms of survival between the combination pemetrexed-carboplatin and pemetrexed alone. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ardizzoni, MD, Principal Investigator — Gruppo Oncologico Italiano di Ricerca Clinica
Locations (21):
- Italy (21):
  - Azienda Ospedaliero-Universitaria Umberto I, Clinica di Oncologia Medica, Ancona
  - Azienda Ospedaliera Ospedali Riuniti di Bergamo, UO di Oncologia Medica, Bergamo
  - Azienda Istituti Ospitalieri di Cremona, UO di Oncologia Medica, Cremona
  - Azienda Sanitaria Ospedaliera S. Croce e Carle, UO di Oncologia Medica, Cuneo
  - Ospedale S. Croce, U.O. di Oncologia Medica, Fano, PU
  - Azienda Ospedaliera Careggi, UO di Oncologia Medica, Florence
  - EO Ospedali Galliera, SC Oncologia Medica, Genova
  - Ospedale Versilia, UO di Oncologia Medica, Lido Di Camaiore, LU
  - USL 6, Presidio Ospedaliero di Livorno, U.O. di Oncologia MedicaAzienda, Livorno
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori-IRST, Oncologia Medica, Meldola, FC
  - Istituto Nazionale Tumori, SC di Oncologia 2, Milan
  - Azienda Ospedaliero-Universitaria di Modena-Policlinico, U.O. di Oncologia Medica ed Ematologia, Modena
  - AO S. Gerardo, Nuovo Ospedale S. Gerardo-settore A, Oncologia Medica, Monza, MI
  - Azienda Ospedaliero-Universitaria di Parma, UOC di Oncologia Medica, Parma
  - Ospedale Silvestrini, S.C. di Oncologia Medica, Perugia
  - Arcispedale Santa Maria Nuova, UO di Oncologia Medica, Reggio Emilia
  - Azienda Ospedaliera S. Camillo-Forlanini, U.O. di Oncologia Medica, Roma
  - Ospedale SS. Annunziata, UO di Oncologia Medica, Sassari
  - Azienda Sanitaria Ospedaliera Molinette, U.O. di Oncologia Medica, Torino
  - P.O. Treviglio-Caravaggio, U.O. di Oncologia Medica, Treviglio, BG
  - Policlinico "G. B. Rossi"-Borgo Roma, U.O. di Oncologia Medica Clinicizzata, Verona

REFERENCES:
- [Derived] van Kruijsdijk RC, Visseren FL, Boni L, Groen HJ, Dingemans AM, Aerts JG, van der Graaf Y, Ardizzoni A, Smit EF. Pemetrexed plus carboplatin versus pemetrexed in pretreated patients with advanced non-squamous non-small-cell lung cancer: treating the right patients based on individualized treatment effect prediction. Ann Oncol. 2016 Jul;27(7):1280-6. doi: 10.1093/annonc/mdw154. Epub 2016 Apr 6. PMID 27052652
- [Derived] Ardizzoni A, Tiseo M, Boni L, Vincent AD, Passalacqua R, Buti S, Amoroso D, Camerini A, Labianca R, Genestreti G, Boni C, Ciuffreda L, Di Costanzo F, de Marinis F, Crino L, Santo A, Pazzola A, Barbieri F, Zilembo N, Colantonio I, Tibaldi C, Mattioli R, Cafferata MA, Camisa R, Smit EF. Pemetrexed versus pemetrexed and carboplatin as second-line chemotherapy in advanced non-small-cell lung cancer: results of the GOIRC 02-2006 randomized phase II study and pooled analysis with the NVALT7 trial. J Clin Oncol. 2012 Dec 20;30(36):4501-7. doi: 10.1200/JCO.2012.43.6758. Epub 2012 Oct 29. PMID 23109689